CLINICAL TRIAL: NCT02381665
Title: INTERFERENTIAL THERAPY IN THE TREATMENT OF CHRONIC CONSTIPATION IN ADULTS: A RANDOMIZED MULTI-CENTER TRIAL
Brief Title: Efficacy of Interferential Therapy in Chronic Constipation (CON-COUR)
Acronym: CON-COUR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-14; 2014-A01359-38 (Registry Identifier: Ansm)
Record Dates: First submitted 2015-02-13; First posted 2015-03-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Constipation Symptoms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Patient enrolled in this group will receive a device for effective interferential current stimulation.
  Interventions: Device: Flexstim IF
- Group B (Placebo Comparator): Patient enrolled in this group will receive a device that does not deliver current stimulation
  Interventions: Device: Flexstim IF faked

INTERVENTIONS:
Device: Flexstim IF — Patient enrolled will receive a device for effective interferential current stimulation
  Arms: Group A
Device: Flexstim IF faked — Patient enrolled will receive a sham device.
  Arms: Group B

SUMMARY:
Chronic constipation is a strong public health problem. Its prevalence is about 15% in Western countries with a significant impact on quality of life and health care costs . Two subtypes of constipation can be identified: slow transit constipation (STC), characterized by impaired propulsion of stool and due to dysfunction of colonic smooth muscle (myopathy) or its innervation (neuropathy), or both; and evacuation disorders, characterized by difficulty or inability with stool expulsion. They include disorders of the anorectal function such as dyssynergic defecation, as well as structural disorders such as rectocele, descending perineum syndrome and rectal prolapse .

The first line therapy of chronic constipation is based on medical treatment combined with laxatives and dietary rules. However, these treatments are often disappointing. In case of failure, few treatment options are currently available. Surgery can sometimes be discussed for intractable chronic constipation. Sub-total colectomy can be proposed in case of STC but is associated with a significant morbidity. In case of pelvic floor disorders, a specific surgical treatment can be indicated. However, surgery is invasive, has a significant morbidity and the results are inconsistent. Recently, some studies have assessed the efficacy of sacral neuromodulation in the treatment of chronic constipation with some success, but this technique is expensive and requires the surgical implantation of a medical device . More recent works, including a randomized trial have showed, in children, the efficacy of interferential current stimulation in the treatment of chronic transit constipation . This treatment is used daily, at home, and uses four adhesive surface electrodes, two abdominal (placed below the costal margin) and two paraspinal (placed between T9 and L2) producing two sinusoidal currents crossing the body, 1 hour per day for 1-3 months. To date, only one open-label study has evaluated this technique in adults and has shown encouraging results in three months with an efficiency on 7/11 patients (63.6%) in the number of stools, severity score of constipation, quality of life's score associated with improved bowel transit time measured by radio-markers.

Interferential therapy is a new treatment that has demonstrated its efficiency in the treatment of chronic constipation in children. Our team has published the first and only pilot study in adults that also demonstrated encouraging results. These data are of particular interest since laxative treatments are often disappointing, are expensive and may have adverse events.

This study would be the first randomized study to evaluate a non-invasive and non-pharmacological treatment of chronic constipation in adults.

If its effectiveness is demonstrated, it will provide, for the first time, a new non-invasive step for patients with laxative treatment failure before considering surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

Subject with a history of chronic constipation defined as:

* two or fewer spontaneous, complete bowel movements per week for a minimum of 6 months before the screening visit*
* or as a sensation of incomplete evacuation or straining during defecation with at least 25% bowel movements*
* Subject with chronic constipation lasting for more than 6 months
* Subject with chronic constipation refractory to medical treatment for at least 3 months (failure or intolerance of medical treatment)
* Subject have to interrupt any laxative treatment but during the study, patients are allowed, in case of absence of bowel movements for 3 or more consecutive days, to take up 15 mg of bisacodyl (Dulcolax, Boerhinger Ingelheim) as rescue medication
* Subjects affiliated to or beneficiary of a social security system
* Subjects who have signed written informed consent

Exclusion Criteria:

* - Minors or pregnant or breast-feeding women
* Subject with chronic constipation secondary to anorectal malformations, to colorectal or anal organic lesions or to a pelvic floor disorder considered by the investigator as necessitating a surgical treatment (rectal prolapse exteriorized, rectocele, enterocele)
* Subjects with current implanted cardiac pacemakers, defibrillators, cardiac pumps, spinal stimulators or other implanted electronic devices
* Subject with chronic constipation secondary to drug, to neurologic, endocrine or metabolic disorders
* Subject with a history of partial colectomy
* Subject with megacolon, megarectum, colonic inertia
* Skin lesions preventing the installation of the electrodes
* Women without effective contraception (hormonal or intra-uterine device)
* Subject misunderstanding the written and spoken French
* Subject participating in another biomedical research protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Number of stool | 8 weeks
  Assessing the short-term efficacy of interferential therapy in adult patients with severe chronic constipation.

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hopitaux De Marseille

REFERENCES:
- [Derived] Vitton V, Mion F, Leroi AM, Brochard C, Coffin B, Zerbib F, Damon H, Melchior C, Duboc H, Queralto M, Baumstarck K. Interferential therapy for chronic constipation in adults: The CON-COUR randomizedcontrolled trial. United European Gastroenterol J. 2023 Apr 25;11(4):337-49. doi: 10.1002/ueg2.12373. Online ahead of print. PMID 37186357
- [Derived] Vitton V, Benezech A, Honore S, Sudour P, Lesavre N, Auquier P, Baumstarck K. CON-COUR study: Interferential therapy in the treatment of chronic constipation in adults: study protocol for a randomized controlled trial. Trials. 2015 May 28;16:234. doi: 10.1186/s13063-015-0752-8. PMID 26012788